CLINICAL TRIAL: NCT02652507
Title: Effect of a Combination of Dexmedetomidine and Ketamine Anesthesia on Upper Airway Morphology in Children
Brief Title: Dexmedetomidine and Ketamine in MRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-0106
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Magnetic Resonance Imaging
Keywords: Sedation; MRI; Dexmedetomidine; Ketamine; General anesthesia; MRI of Brain; MRI of Brain/Spine
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anesthesia for MRI (Other): All patients will receive the same drugs.
  A loading dose of dexmedetomidine of 2 mcg/kg/h over ten minutes followed by a continuous infusion of 2 mcg/kg/h. Bolus dose 2 mg/kg of ketamine will be given after the initial set of research images have been taken.
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — 2 mc/kg/h over ten minutes followed by a continuous infusion of 2 mcg/kg/h
Drug: Ketamine — Bolus dose 2 mg/kg after first set of research images are obtained

SUMMARY:
The purpose of this research study is to examine the effects of two commonly used anesthetic drugs, dexmedetomidine and ketamine, have on the shape and muscle tone of the upper airway in children, adolescents, and young adults.

The results of this study will help in making the best decisions regarding the anesthesia medications used for sedation outside of the operating room.

DETAILED DESCRIPTION:
Upper airway obstruction is a common problem in spontaneously breathing patients under anesthesia. This study is examining the effects of combining dexmedetomidine and ketamine on the muscle tone and airway configuration in children under anesthesia. The hypothesis is adding ketamine to dexmedetomidine will not significantly reduce airway caliber or morphology when compared to previously collected data using dexmedetomidine alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires anesthesia for a MRI scan of the brain or MRI brain/spine
* Patient must be 1 to 18 years of age
* Patients legally authorized representative has given written informed consent to participate in the study

Exclusion Criteria:

* Allergy to dexmedetomidine or ketamine
* History or obstructive sleep apnea
* The patient has a life-threatening medical condition (ASA status 4, 5, or 6)
* The patient is not scheduled to receive anesthesia sedation for the MRI
* Patient has a history or a family history of malignant hyperthermia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Measurement of soft palate under anesthesia | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
  MRI images for research will be taken 4 times during the MRI; estimated additional 6 minutes will be added to the MRI scan
Measurement of base of tongue under anesthesia | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
  MRI images for research will be taken 4 times during the MRI; estimated additional 6 minutes will be added to the MRI scan

SECONDARY OUTCOMES:
Anteroposterior dimension and transverse dimension of soft palate | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
  MRI images for research will be taken 4 times during the MRI; estimated additional 6 minutes will be added to the MRI scan
Anteroposterior dimension and transverse dimension of base of tongue | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
  MRI images for research will be taken 4 times during the MRI; estimated additional 6 minutes will be added to the MRI scan
Patient movement during MRI | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
Episodes of low oxygen saturation | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
Placement of adjunct airway | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
Arterial blood pressure relative to baseline before dexmedetomidine is given | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes
Heart rate relative to baseline before dexmedetomidine is given | Participants will be followed for the duration of the procedure; estimated 60 - 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States